CLINICAL TRIAL: NCT04450147
Title: Efficacy of Tai Chi/Qigong for Subsyndromal Depression and Cognition in Older Age Bipolar Disorder: A Pilot Randomized Controlled Trial With an Active Control
Brief Title: Tai Chi/Qigong for Subsyndromal Depression and Cognition in Older Age Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Soham Rej MD, MSc, Geriatric Psychiatrist, Assistant Professor, Principle Investigator, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-05-2020-1825
Record Dates: First submitted 2020-03-03; First posted 2020-06-29 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2020-11

CONDITIONS: Bipolar Disorder
Keywords: mindfulness; older age bipolar disorder; tai chi; qigong; randomized controlled trial
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tai Chi and Qigong (Experimental): 50mins x 12 weeks of virtually-delivered group tai chi/qigong
  Interventions: Behavioral: Tai Chi/Qigong vs. Walking/Stretching
- Walking and Stretching (Active Comparator): 50mins x 12 weeks of virtually-delivered group walking and stretching
  Interventions: Behavioral: Tai Chi/Qigong vs. Walking/Stretching

INTERVENTIONS:
Behavioral: Tai Chi/Qigong vs. Walking/Stretching — Both interventions can be thought of as a form of movement and exercise.

SUMMARY:
It is expected that by 2030, the percentage of patients with bipolar disorder (BD) in Canada over 60 years of age will exceed 50%. In this population, poor cognition and persistent sub-threshold depressive symptoms are particularly common, difficult to treat, associated with increased mood episodes, and poor daily functioning. Mind-body interventions have increasingly been found to be effective in treating several psychiatric condition including BD. A few pilot studies examining mindfulness-based intervention in younger adult BD have been promising for depressive symptoms, but some pilot research suggest that patients with older age bipolar disorder (OABD) may benefit more from moving mindfulness. The investigators will conduct a 12-week randomized controlled trial to assess whether tai-chi/qigong will be associated with 1) greater reduction in depressive symptoms, and 2) greater improved cognition, in comparison to a light exercise active control condition, 12- and 24-weeks from baseline, in BD patients aged 40+.

ELIGIBILITY:
Inclusion Criteria:

* aged greater than or equal to 40 years
* history of diagnosis of bipolar I or II disorder
* access to a computer with a functioning camera, microphone, and ability to run Zoom software
* English or French speaking
* ability to give informed consent

Exclusion Criteria:

* Young Mania Rating Scale score > 5
* current clinician diagnosis of substance abuse, unless currently in complete remission
* risk of suicide as assessed by a score above 3 on item 10 of Montgomery Asberg Depression Rating Scale
* participation or plan to participate in any other concurrent psychosocial group program during course of study
* unstable psychiatric medication (less than 4-weeks since commencement)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Depression | Baseline, 12-weeks, 24-weeks
  Level of depression as measured by the Montgomery-Asberg Depression Rating Scale, at 12-weeks and 24-weeks post-intervention. Possible score range: 0-60, higher score indicates worse outcome

SECONDARY OUTCOMES:
Change in Processing Speed | Baseline, 12-weeks, 24-weeks
  Processing speed as measured by the Animal Fluency Test at 12-weeks and 24-weeks. Scored by number of animals named, higher score indicates better outcome.

OTHER OUTCOMES:
Change in Quality of Life | Baseline, 12-weeks, 24-weeks
  Quality of life as measured by the Quality of Life in Bipolar Disorder Questionnaire - Short Form, at 12-weeks and 24-weeks post-intervention. Possible score range: 12-60, higher score indicates worse outcome
Change in Daily Functioning | Baseline, 12-weeks, 24-weeks
  Daily functioning as measured by the Functional Assessment Short Test, at 12-weeks and 24-weeks post-intervention. Possible score range: 0-72, higher score indicates worse outcome
Change in Generalized Anxiety | Baseline, 12-weeks, 24-weeks
  Generalized anxiety as measured by the Generalized Anxiety Disorder 7-item scale, at 12-weeks and 24-weeks post-intervention. Possible score range: 0-21, higher score indicates worse outcome
Change in Mindfulness | Baseline, 12-weeks, 24-weeks
  Mindfulness as measured by the Five Factor Mindfulness Questionnaire Short Form at 12-weeks and 24-weeks post-intervention. Possible score range = 49-110, higher score indicates worse outcome
Change in Self-Compassion | Baseline, 12-weeks, 24-weeks
  Self-compassion as measured by the Self Compassion Scale Short Form at 12-weeks and 24-weeks post-intervention. Possible score range: 0-130, higher score indicates worse outcome
Change in Mania | Baseline, 12-weeks, 24-weeks
  Mania as measured by the Young Mania Rating Scale at 12-weeks and 24-weeks post-intervention. Possible score range: 0-60, higher score indicates worse outcome
Change in Self-Reported Depression | Baseline, weekly throughout 12-weeks, 24-weeks
  Level of depression as measured by the Quick Inventory of Depressive Symptomatology - Self Report, at 12-weeks and 24-weeks post-intervention. Possible score range: 0-45, higher score indicates worse outcome
Change in Self-Reported Mania | Baseline, weekly throughout 12-weeks, 24-weeks
  Level of mania as measured by the Altman Self-Rating Mania Scale, at 12-weeks and 24-weeks post-intervention. Possible score range: 0-25, higher score indicates worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Davis Institute, Montreal, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data from the study will be sent to the Global Aging & Geriatric Experiments in Bipolar Disorder Database (GAGE-BD). The objective of GAGE-BD is to gather data from research studies about older adults (age 50+) with bipolar disorder to allow researchers from the Douglas Institute, or other researchers, in Canada, the United States and around the world, to use the database for future research projects exploring possible relationships between age, medical conditions and bipolar symptoms. Following completion of data collection, the data including all outcomes and demographic and health information, anonymized and free of any identifying or personal information, will be sent to Dr. Betsy Wilson (more info on Dr. Wilson further below) via Box (https://case.edu/utech/help/knowledge-base/box/box-information), a secure cloud storage service managed by Case Western University.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available June 2021 (anticipated), and will be kept at GAGE-BD indefinitely.
Access Criteria: All researcher-users involved in GAGE-BD agree not to communicate or transfer data to anyone. They agree not to use the data for a research study that is not approved by the GAGE-BD management or a Research Ethics Board.

REFERENCES:
- [Background] Sajatovic M, Eyler LT, Rej S, Almeida OP, Blumberg HP, Forester BP, Forlenza OV, Gildengers A, Mulsant BH, Strejilevich S, Tsai S, Vieta E, Young RC, Dols A. The Global Aging & Geriatric Experiments in Bipolar Disorder Database (GAGE-BD) project: Understanding older-age bipolar disorder by combining multiple datasets. Bipolar Disord. 2019 Nov;21(7):642-649. doi: 10.1111/bdi.12795. Epub 2019 May 30. PMID 31081573
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/31081573